CLINICAL TRIAL: NCT02843607
Title: Combination of Cryosurgery and NK Immunotherapy for Advanced Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Shenzhen Hank Bioengineering Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NK-kidney
Record Dates: First submitted 2016-07-17; First posted 2016-07-26 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-07

CONDITIONS: Metastatic Renal Cell Cancer
Keywords: Kidney Cancer; Cryosurgery; NK Immunotherapy
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Cryosurgery

ARMS (2):
- Cryosurgery and NK immunotherapy (Experimental): In this group, the patients will receive comprehensive cryosurgery first to destroy all big tumors, then receive multiple NK immunotherapy (intensive treatment: 6 times in first 3 months; then interval treatment: once every 3 months). The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets, circulating tumor cell).
  Interventions: Device: Cryosurgery; Biological: NK immunotherapy
- Cryosurgery (Active Comparator): In this group, the patients will receive comprehensive cryosurgery to destroy all big tumors. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets, circulating tumor cell).
  Interventions: Device: Cryosurgery

INTERVENTIONS:
Device: Cryosurgery — Argon-helium cryosurgical system (percutaneous ablation under CT or ultrasound guidance)
Biological: NK immunotherapy — Natural killer cell (each treatment: about 10 billion cells transfusion in 3 times, i.v.)
  Arms: Cryosurgery and NK immunotherapy

SUMMARY:
The aim of this study is the safety and efficacy of cryosurgery plus NK immunotherapy to advanced kidney cancer.

DETAILED DESCRIPTION:
By enrolling patients with kidney cancer adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of the combined therapy using cryosurgery and nature killer (NK) cells for advanced kidney cancer.

The safety will be evaluated by statistics of adverse reactions. The efficacy will be evaluated according to local relief degree, progress free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* All standard therapies have failed according to NCCN guidelines or the patient refuses standard therapies after cancer recurrence
* Body tumor 1-6, the maximum tumor length < 5 cm
* KPS ≥ 70, lifespan > 6 months
* Platelet count ≥ 80×109/L，white blood cell count ≥ 3×109/L, neutrophil count ≥ 2×109/L, hemoglobin ≥ 80 g/L

Exclusion Criteria:

* Patients with cardiac pacemaker
* Patients with brain metastasis
* Patients with grade 3 hypertension or diabetic complication, severe cardiac and pulmonary dysfunction

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Relief degree | 3 months
  It will be evaluated by the Response Evaluation Criteria in Solid Tumors（RECIST）

SECONDARY OUTCOMES:
Progress free survival（PFS） | 1 year
Overall survival（OS） | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Guifeng Liu, PhD, Principal Investigator — Fuda Cancer Hospital, Guangzhou
Locations (1):
- Cancer Institute in Fuda cancer hospital, Guangzhou, Guangdong, China